CLINICAL TRIAL: NCT06470438
Title: A Phase 1, First-in-Human, Dose Escalation Study of JNJ-88998377 in Participants With Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: A Study of JNJ-88998377 for Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 88998377LYM1001; 88998377LYM1001 (Other: Janssen Research & Development, LLC); 2023-509258-71-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin; Refractory B-Cell NHL; Relapsed B-cell NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A: Dose Escalation (Experimental): Participants will receive JNJ-88998377 at a selected starting dose. Subsequent dose levels and schedules will be selected based on the review of all available data to establish recommended Phase 2 dose (RP2D).
  Interventions: Drug: JNJ-88998377
- Part B: Dose Expansion (Experimental): Participants will receive JNJ-88998377 at RP2D determined in Part A. Additional expansion cohort(s) may be added with a lower RP2D(s), or different dose schedule(s) based on all available data.
  Interventions: Drug: JNJ-88998377

INTERVENTIONS:
Drug: JNJ-88998377 — JNJ-88998377 will be administered.

SUMMARY:
The main purpose of this study is to characterize safety and to determine the recommended phase 2 dose (RP2D) for JNJ-88998377 (Part A: Dose Escalation), to further assess the safety of JNJ-88998377 at the RP2D (Part B: Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

* Participants have histologically or cytologically confirmed B-cell non-Hodgkin's Lymphoma (NHL) according to the 2022 World Health Organization (WHO) classification with relapsed or refractory disease
* Participants have measurable disease or meet all requirements for adequate response assessment as defined by the appropriate disease response criteria at screening
* Participants have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants have a life expectancy of greater than or equal to (>=) 12 weeks
* Be willing and able to adhere to the lifestyle restrictions specified in the protocol

Exclusion Criteria:

* Participant with active or prior history of B-cell NHL involving the central nervous system (CNS) and leptomeningeal involvement
* History of malignancy (other than the disease under study in the cohort to which the participant is assigned) within 1 year prior to the first administration of study treatment.
* For Part A and B: Participant having known allergies, hypersensitivity, or intolerance to the excipients of JNJ-88998377
* Participant had major surgery or had significant traumatic injury within 30 days before first dose of study treatment or has not recovered from surgery and must not have major surgery planned during the time the participant is receiving study treatment
* Participant received an autologous stem cell transplant less than or equal to (<=) 3 months before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2028-10-18 (Estimated)

PRIMARY OUTCOMES:
Parts A and B: Number of Participants with Adverse Events (AEs) | Upto 3 years 4 months
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical (investigational or non-investigational) product. It does not necessarily have a causal relationship with the investigational product.
Part A: Number of Participants with Dose Limiting Toxicity (DLTs) | Cycle 1 (21 days)
  Number of participant with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematological or hematological toxicity.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-88998377 | Up to first 12 weeks
  Plasma concentration of oral dose of JNJ-88998377 will be assessed.
Area Under the Plasma Concentration Versus Time Curve During A Dosing Interval (τ) At Steady-State of JNJ-88998377 | Up to first 12 weeks
  Area under the plasma concentration versus time curve during a dosing interval (τ) at steady-state concentration of JNJ-88998377 will be reported.
Maximum Plasma Concentration (Cmax) of JNJ-88998377 | Up to first 12 weeks
  Cmax of JNJ-88998377 will be reported.
Minimum Plasma Drug Concentration (Cmin) of JNJ-88998377 | Up to first 12 weeks
  Cmin of JNJ-88998377 will be reported.
Percentage of Participants With Overall Response (OR) | Up to 3 years 4 months
  OR is defined as the percentage of participants who have a best response of partial response (PR) or better per investigator assessment according to disease-specific response criteria.
Time to Response (TTR) | From first dose of study treatment until first response of PR or better (up to 3 years and 4 months)
  TTR is defined for participants who achieved a response of PR or better as the time from the first dose of study treatment to the first response of PR or better per investigator assessment according to disease-specific response criteria.
Duration of Response (DOR) | From date of documentation of first response of PR or better until progressive disease or death (up to 3 years and 4 months)
  DOR is defined for participants who achieved a response of PR or better as the time between the date of initial documentation of first response of PR or better to the date of first documented evidence of progressive disease or death.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (19):
- China (5):
  - Beijing Cancer Hospital, Beijing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
- A O U Sant Orsola Malpighi, Bologna, Italy
- Japan (3):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (3):
  - Pratia Onkologia Katowice, Katowice
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Klinika Hematologii i Transplantacji Szpiku, Kielce
  - Aidport Sp z o o, Skorzewo
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (3):
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Koc University Medical Faculty, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency